CLINICAL TRIAL: NCT03649672
Title: The Validity and Tolerability of Awake Calibration of the TOF Watch SX® Monitor: An Interventional Prospective Single Two-center Study
Brief Title: The Validity and Tolerability of Awake Calibration of the TOF Watch SX Monitor
Acronym: CaliRev
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid Crisis recruitment was stopped.
Sponsor: Christoph Czarnetzki (Other)
Collaborators: Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Christoph Czarnetzki, MD, MBA, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CaliRev
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Neuromuscular Blockade
Keywords: Tof Watch, rocuronium

STUDY DESIGN:
Intervention Model Description: Neuromuscular monitoring by TOF Watch SX on the dominant and on the non dominant arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Awake calibration (Experimental): The dominant arm of the patient
  Interventions: Device: TOF Watch SX
- Asleep calibration (Active Comparator): The non dominant arm of the patient
  Interventions: Device: TOF Watch SX

INTERVENTIONS:
Device: TOF Watch SX — Neuromuscular monitoring via the TOF Watch SX device

SUMMARY:
Neuromuscular blocking agents (NMBAs) are frequently used in anesthesia and quantitative monitoring of neuromuscular block is standard care. Normally the calibration of the neuromuscular monitor is done after anesthesia induction to avoid patient discomfort. Under certain circumstances there is no time for the calibration process. In the so-called rapid sequence induction (RSI) the neuromuscular blocking agent has to be injected immediately after the induction agent. As the neuromuscular monitor cannot be calibrated, precise neuromuscular monitoring is not possible, and this is of particular disadvantage, when high doses of non-depolarizing neuromuscular blockers are injected to fasten the onset of neuromuscular block. The primary objective is to validate the measurements of the TOF Watch SX® monitor calibrated in awake patients by comparing them with the measurements obtained with the TOF Watch SX® monitor calibrated after anesthesia induction (Gold standard).

The secondary objective is to evaluate the tolerability of the awake calibration process of the TOF Watch SX® monitor.

DETAILED DESCRIPTION:
Neuromuscular function will be assessed by acceleromyography of the adductor pollicis with a TOF-Watch SX® monitor on both arms. By randomization it will be chosen on which arm the awake calibration will be done. 5 minutes before the awake calibration process the patients will receive 0.2 µg/kg of sufentanil intravenously. Immediately after the end of the calibration process the patients will rate the pain of the calibration process on a visual analog scale from 0 to 10. Anesthesia will then be induced and immediately at loss of consciousness continuous TOF stimulation will be continued every 12s. Then the calibration process on the other arm will be started, followed by continuous TOF stimulation. After having obtained stable baseline measurements with the TOF-Watch SX® monitor, a bolus dose of rocuronium 0.6 mg kg-1 will be administered intravenously. The trachea will be intubated when full neuromuscular block is reached. No additional rocuronium will be given. Both neuromuscular monitors will be linked via a fiber-optic (TOF-Link®) cable with UBS port to a laptop. Specific software will be used to record the measurements (TOF watch SX® monitor, version 2.2). Neuromuscular monitoring will be continued until a normalized TOF ratio of 0.9 has been obtained on both arms. The onset of neuromuscular block and its spontaneous recovery will be recorded and the results obtained on each arm will be compared. Every patient is his own control.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II
* patients undergoing elective surgery lasting at least 60 minutes under general anesthesia requiring neuromuscular blockade using rocuronium bromide for endotracheal intubation

Exclusion Criteria:

* Patient with a history of allergy or hypersensitivity to rocuronium.
* Patients with neuromuscular disease
* Patients with preoperative medications known to influence neuromuscular function (for instance aminoglycosides, phenytoin, lidocaine)
* Patients with electrolyte abnormalities (for instance, hypermagnesemia)
* Patients with a body mass index <19 or >30 kg m2
* Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial
* Patients undergoing interventions that need a continuous deep neuromuscular block
* Pregnant or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Total recovery time | during the duration of the general anesthesia
  Total duration of the neuromuscular block defined as the time in minutes from start of injection of rocuronium until a normalized TOF ratio of 90%

SECONDARY OUTCOMES:
Onset time | during the duration of the general anesthesia
  The time in seconds from start of injection of rocuronium until 95% depression of the first twitch (T1) of the TOF
Dur TOFc1 | during the duration of the general anesthesia
  Time in minutes from administration of rocuronium to emergence of the 1st twitch of the TOF
Dur TOF 25% | during the duration of the general anesthesia
  Time in minutes from administration of rocuronium to emergence of a TOF ratio of 25%
Dur TOF 50% | during the duration of the general anesthesia
  Time in minutes from administration of rocuronium to emergence of a TOF ratio of 50%
Dur TOF 75% | during the duration of the general anesthesia
  Time in minutes from administration of rocuronium to emergence of a TOF ratio of 75%
TOF pain: VAS | before inductin of general anesthesia
  The pain experienced during the calibration process evaluated by a visual analogue scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, Study Chair — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - University Hospital of Geneva, Anesthesia Department, Geneva, Canton of Geneva
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino